CLINICAL TRIAL: NCT02090465
Title: Assessment of Treatment Success and Quality of Life in Patients With Actinic Keratoses Under Therapy With Ingenol Mebutate (Picato) in a Period of 8 Weeks.
Brief Title: Assessment of Treatment Success and Quality of Life in Patients With Actinic Keratoses Under Therapy With Ingenol Mebutate in a Period of 8 Weeks
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: DE-Picato NIS-2013
Record Dates: First submitted 2014-03-12; First posted 2014-03-18 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all eligible patients: Treatment with Picato according to Summary of Product Characteristics (SmPC)
  Interventions: Drug: Ingenol Mebutate

INTERVENTIONS:
Drug: Ingenol Mebutate — No intervention: observation of routine use of Picato®
  Other Names: Picato®

SUMMARY:
Assessment of treatment success and quality of life in patients with actinic keratoses under therapy with Ingenol Mebutate (Picato) in a period of 8 weeks.

DETAILED DESCRIPTION:
Non-interventional (observational) study (NIS), non-controlled, prospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

• Non-hyperkeratotic, non-hypertrophic actinic keratoses where treatment with Picato® is indicated and the treatment is intended by physicians.

Exclusion Criteria:

* Preceding use of Picato® on the area planned for treatment
* Any other specific local treatment of actinic keratoses on the area planned for treatment during the last 8 weeks
* Melanoma, squamous cell carcinoma or spinalioma on the area planned for treatment
* Open wounds on the area planned for treatment
* Contraindications according to prescribing information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with actinic keratosis contacting their dermatologist
Sampling Method: Non-Probability Sample
Enrollment: 840 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Actinic keratosis | 8 weeks
  Documentation of the course of actinic keratoses and skin findings during ambulant routine use of Picato®
Skindex-16 | 8 weeks
  Patient' s quality of life during ambulant routine use of Picato®
Dosage of Picato® | 8 weeks
  Prescribed and applied dosages and adherence during ambulant routine use of Picato®

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Diepgen, Prof. Dr. med., Principal Investigator — University Hospital Heidelberg
Locations (1):
- Universitätsklinikum Heidelberg/Klinische Sozialmedizin, Heidelberg, Germany